CLINICAL TRIAL: NCT05227040
Title: Effect of the Nintendo Ring Fit Adventure Exergame on Running Completion Time and Psychological Factors Among University Students Engaging in Distance Learning During the COVID-19 Pandemic: A Randomized Prospective Study
Brief Title: Effect of the Nintendo Ring Fit Adventure Exergame on Running Completion Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, WU, YI - SYUAN, Principal Investigator, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NDMC_Chulab_002
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Sleep Quality; Mood Disorders
Keywords: Exergaming; Cardiac force index; Running; Physical activity; Sleep quality; Mood disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mood Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nintendo Ring Fit Adventure Exergame Group (Experimental): Participants in the RFA group were required to exercise for 30 minutes three times per week (in adventure mode) for 4 weeks. The initial exercise intensity was set according to the instructions given by the virtual coach during the first game and was gradually adjusted according to the game instructions. The research continued to track the RFA group subjects and continued to encourage the completion of 4 weeks of physical activity training.
  Interventions: Device: Nintendo Ring Fit Adventure Exergame
- Control group (No Intervention)

INTERVENTIONS:
Device: Nintendo Ring Fit Adventure Exergame — Participants in the RFA group were required to exercise for 30 minutes three times per week (in adventure mode) for 4 weeks. The initial exercise intensity was set according to the instructions given by the virtual coach during the first game and was gradually adjusted according to the game instructions. The research continued to track the RFA group subjects and continued to encourage the completion of 4 weeks of physical activity training.
  Arms: Nintendo Ring Fit Adventure Exergame Group

SUMMARY:
The coronavirus disease 2019 (COVID-19) outbreak has not only changed the lifestyles of people globally but has also resulted in other challenges, such as the requirement of self-isolation and distance learning. The COVID-19 pandemic has resulted in an inability to go out to exercise and a reduction in movement, so the demand for exercise at home has increased. To investigate the relationships between a Nintendo Ring Fit Adventure (RFA) intervention and improvements in running time, cardiac force index (CFI), centimeters per beat (CMPB), sleep quality, and mood disorders.

DETAILED DESCRIPTION:
In this study, a pre-test-post-test control group design was used to collect data from healthy populations in the northern region. The intervention groups were simply randomly assigned to investigate the cardiac force index, sleep quality and mood disorders before and after 4 weeks of Ring Fit Adventure intervention. The study will use the wearable Medtronic ZephyrTM BioHarness 3.0 and Q-Band HR3 (Q-69HR) bracelet. The device is used for physiological parameter collection. Heart rate, acceleration, activity acceleration, activity volume, CFI were recorded during a 1600 m run for pre-post-test.

In this study, ZephyrTM BioHarness 3.0 and a Q-Band HR3 (Q-69HR) bracelet were used to collect as physiological parameters. Heart rate, acceleration, activity, cardio index and cardio force ratio were recorded before and after 1600 meters.

In order to know whether there are relevant influencing factors for the mental strength indicators in this study, the gender, age, height, weight, neck circumference, waist circumference, hip circumference, smoking and drinking habits, and family medical history of the case will be recorded, and the GPS track during running will be recorded before and after each running. Time, distance, ambient temperature and humidity, weight, neck circumference, waist circumference, hip circumference, blood pressure, blood oxygen, heart rate, etc., and analyze the relationship between parameters. The above cases are measured and recorded every time they run. This is a longitudinal cohort study. The statistics will be repeated variable analysis and generalized linear model, etc., to explore the norm estimation of CFI in different ages and genders.

Before using Microsoft Office 365 Excel for data archiving and analytical processing, please study the data, including the compilation of Zephyr BioHarness data and the calculation of the heart rate index. According to statistical analysis methods, in descriptive statistical analysis, categorical data are presented in numbers and percentages, while continuous data are presented in mean and standard deviation presentations.

Inference statistics will be analyzed using paired t-tests, ANOVA, and generalized linear models to analyze cardiac force before and after the intervention. If the data were not normally distributed, the analysis was performed using the Wilcoxon signed-rank test. The significance level for this study was set at α = 0.05. All analytical data pipelines will use IBM SPSS Statistics version 26. The data has been delinked when the case is received, and personal data cannot be recalled in any way. The received data is stored in a server with account and password control.

ELIGIBILITY:
Inclusion Criteria:

* students who were over 20 years old and did not have chronic diseases;
* students who were able to complete the 1600-meter outdoor run before and after the intervention;
* students who understood and agreed with the research purpose and signed the consent form.

Exclusion Criteria:

* chronic diseases or medications prescribed for over 6 months;
* restricted movement or failure to complete the 1600-meter run before and/or after the intervention
* wearable devices that were not worn well or inability to calculate the cardiac force index (CFI).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Running Completion Time | 4 week
  Investigators researched to use a 1600-meter running for testing.

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu YS, Wang WY, Chan TC, Chiu YL, Lin HC, Chang YT, Wu HY, Liu TC, Chuang YC, Wu J, Chang WY, Sun CA, Lin MC, Tseng VS, Hu JM, Li YK, Hsiao PJ, Chen CW, Kao HY, Lee CC, Hsieh CB, Wang CH, Chu CM. Effect of the Nintendo Ring Fit Adventure Exergame on Running Completion Time and Psychological Factors Among University Students Engaging in Distance Learning During the COVID-19 Pandemic: Randomized Controlled Trial. JMIR Serious Games. 2022 Mar 22;10(1):e35040. doi: 10.2196/35040. PMID 35315780